CLINICAL TRIAL: NCT02066831
Title: Diabetes Coaching Study
Acronym: DCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West German Center of Diabetes and Health (Other)
Collaborators: German Institute for Telemedicine and Health Promotion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DCS
Record Dates: First submitted 2014-02-17; First posted 2014-02-20 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemedical Coaching (Experimental): Patients will receive telemedical devices i.e. for the measurement of blood glucose, weight and physical activity. These devices will transfer the data to a data collector with a SIM card which sends the data to a data portal, which can be monitored by the participant and the coach. Health coaches which will have close phone contact to patients, supporting them to reduce weight and increase physical activity. In the first 12 weeks, patients will follow a formula diet (Almased) to achieve an initial weight reduction.
  Interventions: Behavioral: Telemedical coaching; Other: Telemedicine
- Telemedicine (Active Comparator): Patients will receive telemedical devices i.e. for the measurement of blood glucose, weight and physical activity. These devices will transfer the data to a data collector with a SIM card which sends the data to a data portal which can be monitored by the participant.
  Interventions: Behavioral: Telemedical coaching

INTERVENTIONS:
Behavioral: Telemedical coaching
Other: Telemedicine
  Arms: Telemedical Coaching

SUMMARY:
The purpose of the study is to compare the effect of telemedical coaching versus telemedical control on HbA1c, weight, BMI, blood pressure, blood lipids, medication, nutrition, physical activity and quality of life in type 2 diabetes patients with poor glycaemic control.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus
* hemoglobin A1c (HbA1c) >7.5%
* at leat two different antidiabetic drugs
* body mass index >27kg/m2

Exclusion Criteria:

* acute infections
* diagnosed chronic diseases other than type 2 diabetes and hypertension, e.g. cancer, chronic obstructive pulmonary disease (COPD), asthma, dementia, chronic gut diseases, psychoses, liver cirrhosis, (macro-) nephropathy, kidney insufficiency with glomerular filtration rate (eGFR) < 30ml / min / 1.73 m2
* acute chemotherapy or chronic cortisol treatment
* smoking cessation for less than 3 months and or planned smoking cessation during study
* known intolerance of any ingredient of Almased (especially soy protein)
* pregnancy or breast feeding, lack of contraception (women)
* other study participation in the last 6 months prior to study start

Ages: 25 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2014-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
HbA1c | 12 months
  Difference in HbA1c (at end of study vs. baseline) between the groups

SECONDARY OUTCOMES:
weight | 12 months
  Difference in weight (at end of study vs. baseline) between the groups
antidiabetic medication | 12 months
  Difference in antidiabetic medication (at end of study vs. baseline) between the groups
Cardiovascular risk parameters (blood pressure, blood lipids) | 12 months
  Difference in cardiovascular risk parameters (i.e. blood pressure, blood lipids) (at end of study vs. baseline) between the groups
physical activity (step count) | 12 months
  Difference in physical activity (at end of study vs. baseline) between the groups
nutrition | 12 months
  Difference in nutrition (at end of study vs. baseline) between the groups
quality of life | 12 months
  Difference in quality of life (at end of study vs. baseline) between the groups

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Martin, MD, Principal Investigator — West German Center of Diabetes and Health
Locations (1):
- West-German Center of Diabetes and Health, Düsseldorf, Germany

REFERENCES:
- [Derived] Kempf K, Altpeter B, Berger J, Reuss O, Fuchs M, Schneider M, Gartner B, Niedermeier K, Martin S. Efficacy of the Telemedical Lifestyle intervention Program TeLiPro in Advanced Stages of Type 2 Diabetes: A Randomized Controlled Trial. Diabetes Care. 2017 Jul;40(7):863-871. doi: 10.2337/dc17-0303. Epub 2017 May 12. PMID 28500214
- See also: Homepage — http://www.vkkd-kliniken.de